CLINICAL TRIAL: NCT02339077
Title: Group B Streptococcus (GBS) Associated Stillbirths in a High Burden Setting
Acronym: Stillborn
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Farzanah Laher, Dr, University of Witwatersrand, South Africa
Other Study IDs: V98_27OBTP
Record Dates: First submitted 2014-08-11; First posted 2015-01-15 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2018-09

CONDITIONS: Stillbirth
Keywords: Group B Streptococcus, stillborn
MeSH Terms: conditions — Stillbirth

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Cord blood Placenta skin swab from fetus Gastric/ tracheal aspirate
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a descriptive study to determine the role of fetal GBS disease as a cause for stillbirths

DETAILED DESCRIPTION:
A prospective, descriptive study will be undertaken involving mothers who have a stillbirth at Chris Hani Baragwanath Academic Hospital (CHBAH), a secondary-tertiary care hospital, from 2014 up until 2016.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women delivering a stillbirth at CHBAH
* Participants aged ≥18 years
* Able to understand and comply with planned study procedures
* Provides written informed consent (either generic ICF or V98_28OBTP)

Exclusion Criteria:

* Refuses to consent to study participation

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Stillborn infants (gestational age >= 28 weeks gestation) born at CHBAH
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determine the number of stillbirths who have GBS isolated from cord blood, gastric aspirates, placenta and/ or skin swabs | Birth

SECONDARY OUTCOMES:
Number of stillbirths occurring at CHBAH, and identify potential causes of the stillbirths (maternal and obstetric risk factors) | Birth
  To determine the epidemiology of stillbirths, including identification of maternal risk-factors
Number of stillbirths related to a probable Infectious cause | Birth
  To determine the proportion of stillbirths that are associated with common fetal in-utero infections including; Syphilis (Treponema pallidum), Klebsiella sp, E. Coli

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - Respiratory and Meningeal Pathogen Research Unit, Johannesburg, Gauteng
  - Chris Hani Baragwanath Academic Hospital, Johannesburg, Gauteng